CLINICAL TRIAL: NCT01837771
Title: Uni- or Biventricular Pacing and Diaphragmatic Stimulation for Severe Heart Failure (Epiphrenic III Pilot Trial)
Brief Title: Epiphrenic III Pilot Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Luzerner Kantonsspital (Other)
Responsible Party: Principal Investigator, Prof. Paul Erne, Head of Department of Cardiology, Luzerner Kantonsspital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 13008
Record Dates: First submitted 2013-04-16; First posted 2013-04-23 (Estimated); Last update posted 2013-04-23 (Estimated); Status verified 2013-04

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

ARMS (2):
- Diaphragmatic stimulation (Active Comparator): Diaphragmatic stimulation via electrode for 4 weeks
  Interventions: Device: Diaphragmatic stimulation
- No intervention (No Intervention)

INTERVENTIONS:
Device: Diaphragmatic stimulation
  Arms: Diaphragmatic stimulation

SUMMARY:
The Epiphrenic III Pilot Trial investigates whether a diaphragmatic stimulation by interventionally placed electrodes may improve heart function, symptoms and functional capacity in patients with severe heart failure.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic heart failure (NYHA functional classes II, III or IV)
* Reduced left ventricular ejection fraction (LVEF) <35%
* Guideline-recommended drug therapy

Exclusion Criteria:

* Patient refuses study participation
* Life expectancy presumably <1 year
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2013-04; Primary Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Left ventricular ejection fraction | Four weeks
NYHA functional class | Four weeks

SECONDARY OUTCOMES:
Brain natriuretic peptide (BNP) | Four weeks
6-minutes walking test | Four weeks

CONTACTS AND LOCATIONS:
Overall Officials: Paul Erne, MD, Principal Investigator — Luzerner Kantonsspital
Locations (1):
- Luzerner Kantonsspital, Lucerne, Canton of Lucerne, Switzerland